CLINICAL TRIAL: NCT07251179
Title: Characterization of Autoreactive b Lymphocytes in Autoimmune Diseases and Immune Deficiencies
Acronym: AutoB-Tetramer
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9942
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus; Systemic Scleroderma; ANCA-associated Vasculitis; Antiphospholipid Syndrome; Primary Immunodeficiencies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Antiphospholipid Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Systemic lupus erythematosus
  Interventions: Biological: blood draw
- Systemic scleroderma
  Interventions: Biological: blood draw
- ANCA-associated vasculitis
  Interventions: Biological: blood draw
- Antiphospholipid syndrome
  Interventions: Biological: blood draw
- Primary immunodeficiencies
  Interventions: Biological: blood draw

INTERVENTIONS:
Biological: blood draw — blood draw

SUMMARY:
Autoimmune diseases (AID), whether systemic or organ-specific, affect approximately one in ten people, and their prevalence continues to increase. Many AIDs are linked to the emergence of autoreactive B cells (BCs) directed against components of the self. In healthy individuals, these autoreactive B cells are counter-selected or regulated before reaching the antibody-secreting cell compartment. However, in predisposed individuals, a breakdown in B cell tolerance can occur, leading to the formation of autoantibodies with devastating consequences, such as the emergence of systemic lupus erythematosus (SLE), rheumatoid arthritis, and vasculitis. B-cell depletion is often beneficial in these patients, but paradoxically, therapies targeting B cells are not always effective. Furthermore, B cell depletion via LB-specific antibodies (anti-CD20) or treatment with CD19 chimeric antigen receptor T cells (CAR T) leads to complete and prolonged depression of the entire B compartment without targeting the LB population responsible for the onset of the disease. To date, two pitfalls in studies of human autoreactive LBs often complicate the interpretation of results:

i) the difficulty of identifying autoreactive LBs among all LBs, ii) demonstrating the pathogenicity of autoreactive B lymphocytes when they can be identified individually. We propose to quantify and phenotype these autoreactive/pathogenic B cells using high-throughput flow cytometry in several clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70
* Patients for whom at least one of the following conditions has been confirmed:
* Systemic lupus erythematosus meeting the 2019 ACR/EULAR classification criteria.
* Systemic scleroderma meeting the 2013 ACR/EULAR classification criteria. ANCA-associated vasculitis according to the 2022 EULAR/ACR classification criteria.
* Antiphospholipid syndrome according to the 2023 ACR/EULAR criteria.
* Primary immunodeficiencies according to IUIS criteria.
* Patients capable of understanding the objectives of the research.
* Patients affiliated with a social security health insurance scheme (beneficiary or dependant).
* Patients who have signed and dated the informed consent form for non-identifying genetic testing.

Exclusion Criteria:

* Patient refusing to participate in the study
* Patient in a period of exclusion (determined by a previous or ongoing study) Inability to provide the subject with informed consent (in an emergency or immediate life-threatening situation, difficulties in understanding the subject, etc.)
* Patient under legal protection
* Patient under guardianship or conservatorship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hôpitaux Universitaires de Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Study of the percentage of autoreactive LB / tetrameric LB+ | inclusion visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France